CLINICAL TRIAL: NCT02836951
Title: Rapid Chemical Diagnostics of Brain Injuries
Brief Title: Rapid Diagnostics for Traumatic Brain Injury (TBI)
Status: Completed | Type: Observational
Sponsor: Medicortex Finland Oy (Industry)
Collaborators: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: T129/2016
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood, urine, and saliva.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient: This group consists of patients that are hospitalized due to a head injury. Samples of blood, urine and plasma will taken from these subjects and the fluids will be analyzed for novel biomarkers using a biochemical assay.
  Interventions: Other: Withdrawal of blood
- Healthy controls: This group consists of healthy volunteers. Samples of blood, urine and plasma will taken from these subjects and the fluids will be analyzed for novel biomarkers using a biochemical assay.
  Interventions: Other: Withdrawal of blood

INTERVENTIONS:
Other: Withdrawal of blood — Withdrawal of blood

SUMMARY:
Novel biomarkers of traumatic brain injury (TBI) have been discovered in laboratory animal models. The objective of this study is to find whether similar markers are detectable in the body fluids of human subjects that have sustained a TBI.

DETAILED DESCRIPTION:
Staff of the Neurosurgical ward is asked to report to the study coordinator all patients who are hospitalized due to a suspected brain injury. After an informed consent is received, the patient has been enrolled in the study and sample collection can be started. Plasma samples are taken by the TYKSlab personnel, and the other samples by the nurses in the Neurosurgical ward. The sampling will be organized so that all the samples from a patient are preferably collected at one event. Samples will stored in the TYKSlab at the temperature of -70 °C. Collection of a sufficient number of samples (patients) will take a few months, and subsequent analysis by the Sponsor a few months. All the activities will be done during the years 2016 to 2017.

When the samples of 24 subjects have been collected, they will be transferred to the Sponsor who will ship them further to the sub-contractors. The results received from the research laboratories will be evaluated by the scientist team at Medicortex Finland Oy. The results will be published in a scientific journal, when considered to be of high enough quality and impact.

ELIGIBILITY:
Inclusion Criteria:

* Patient is hospitalized because of a head trauma and suspected TBI.
* Age 18 or above. The subject (including the control subjects) must be an independent adult who is not under guardianship.
* The patient, or the next of kin in the case of an incompetent person, has signed the Informed consent. This concerns the control subjects, too.
* The samples can be collected during regular office hours.
* The patient needs lumbar puncture for treatment reasons. This is not a limiting criterion however. If it is difficult to find an adequate number of patients for lumbar puncture, CSF samples of some patients can be omitted after the study coordinator's consideration.

Exclusion Criteria:

* The subject has been found positive for HIV or hepatitis-B in the involved laboratory studies.
* The subject has a chronic mental disorder which is mentioned on the sickness insurance card.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will include patients that are hospitalized due to a suspected traumatic brain injury. Identical number of healthy volunteers will serve as controls.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Presence of lectin-complexes in patients with TBI | Two years
  There is a difference in the intensity of immuno-fluorescence readings between TBI patients and healthy controls. Different lectin bound complexes will be studied in body fluid samples collected from the patients (the trial is not following the patients nor is it intended to evaluate clinical outcome).
Characterization of molecule structure of lectin-complexes | Two years
  Molecular characterization of lectin-complexes by HPLC (high performance liquid chromatography) and MS (mass spectrometry) analysis. Samples retrieved from the patients are being analyzed comparing head injured to healthy controls. No follow-up of the patients and no clinical evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Jaakko Rinne, Professor, Principal Investigator — University of Turku
Locations (1):
- Turku University Hospital (Tyks), Turku, Finland